CLINICAL TRIAL: NCT00900627
Title: A Phase I/II Multi-centre Study of AZD8931 in Combination With Weekly Paclitaxel to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy in Patients With Advanced Solid Tumours and in a Selected Population With Low HER2-expressing Locally Recurrent and/or Metastatic Breast Cancer
Brief Title: Phase I/II AZD8931/Paclitaxel in Treatment of Advanced Solid Tumours (Phase I) and Advanced Breast Cancer (Phase II)
Acronym: THYME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0102C00003
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Neoplasms; Breast Neoplasms; Breast Cancer
Keywords: Cancer; Tumour; Breast cancer; Metastatic; Secondary
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — AZD 8931; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AZD8931 plus Paclitaxel
  Interventions: Drug: AZD8931; Drug: Paclitaxel
- 2 (Placebo Comparator): Placebo plus Paclitaxel
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: AZD8931 — Tablet Oral bid
  Arms: 1
Drug: Paclitaxel — IV once weekly for 3 weeks followed by a week off (repeated cycles)
  Other Names: Taxol
Drug: Placebo — Oral bid (twice daily)
  Arms: 2

SUMMARY:
The main purpose of this study is to determine if AZD8931 can improve the efficacy of standard chemotherapy for the treatment of advanced breast cancer. This study will be conducted in 2 parts: the first part (phase I) will determine a dose of AZD8931 that can be safely administered with paclitaxel chemotherapy. The second part (phase II) will determine the efficacy and safety of AZD8931 in combination with paclitaxel chemotherapy in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male/ female with solid, malignant tumour which is unresponsive to standard therapies (Phase I). Female patients with advanced breast cancer with low HER2 expression (Phase II)
* Suitable for paclitaxel chemotherapy
* Life expectancy more than 12 weeks

Exclusion Criteria:

* Inadequate kidney, liver, heart, gastric, lung or eye function
* Hypersensitive to paclitaxel
* No symptomatic uncontrolled brain metastases
* Previous taxane chemotherapy within 12 months (Phase II)

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2009-06; Primary Completion 2012-04 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Serban Ghiorghiu, Study Director — AstraZeneca; Professor Jose Baselga, Principal Investigator — Vall d'Hebron University Hospital
Locations (38):
- Belgium (4):
  - Research Site, Brussels (Jette)
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Sint-Niklaas
- Research Site, São Paulo, Brazil
- Bulgaria (4):
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Vratsa
- Canada (3):
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
- Czechia (6):
  - Research Site, Brno
  - Research Site, Jičín
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Praha 4 - Krc
  - Research Site, Znojmo
- Research Site, Villejuif, France
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Szeged
- Italy (3):
  - Research Site, Lido di Camaiore
  - Research Site, Modena
  - Research Site, Treviglio
- Research Site, Panama City, Panama
- Research Site, Lima, Peru
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
- Research Site, Uppsala, Sweden
- Research Site, Chur, Switzerland
- United Kingdom (5):
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I: 20 patients enrolled, 6 to AZD8931 160mg, 2 to AZD8931 120 mg, 6 to AZD8931 80 mg and 6 to AZD8931 40mg. Phase II: 305 enrolled, 190 randomised, 94 and 96 allocated to AZD8931 40mg + Paclitaxel and Placebo + Paclitaxel respectively. Enrolled patients differs slightly from protocol as focus was on achieving number to be randomised.
Groups:
- AZD8931 160 mg bd: Part A: AZD8931 160mg (bd) plus weekly paclitaxel of 90mg/m2 on days 1, 8 and 15 of each 28 day cycle
- AZD8931 120 mg bd: Part A: AZD8931 120mg (bd) plus weekly paclitaxel of 90mg/m2 on days 1, 8 and 15 of each 28 day cycle
- AZD8931 80 mg bd: Part A: AZD8931 80mg (bd) plus weekly paclitaxel of 90mg/m2 on days 1, 8 and 15 of each 28 day cycle
- AZD8931 40 mg bd: Part A: AZD8931 40mg (bd) plus weekly paclitaxel of 90mg/m2 on days 1, 8 and 15 of each 28 day cycle
- AZD8931 40MG bd + Paclitaxel: Part B: AZD8931 40mg (bd) plus weekly paclitaxel of 90mg/m2 on days 1, 8 and 15 of each 28 day cycle
- Placebo + Paclitaxel: Part B: Placebo (bd) plus weekly paclitaxel of 90mg/m2 on days 1, 8 and 15 of each 28 day cycle
Period: Overall Study
Arm/Group | AZD8931 160 mg bd | AZD8931 120 mg bd | AZD8931 80 mg bd | AZD8931 40 mg bd | AZD8931 40MG bd + Paclitaxel | Placebo + Paclitaxel
Started | 6 | 2 | 6 | 6 | 94 (The values under 'Not Completed' are based on the time of the primary analysis) | 96 (The values under 'Not Completed' are based on the time of the primary analysis)
Completed | 0 (No set completion, patients were to remain in study until withdrawn) | 0 (No set completion, patients were to remain in study until withdrawn) | 0 (No set completion, patients were to remain in study until withdrawn) | 0 (No set completion, patients were to remain in study until withdrawn) | 65 (No set completion, pts were to remain in study until withdrawn) | 70 (No set completion, patients were to remain in study until withdrawn)
Not Completed | 6 | 2 | 6 | 6 | 29 | 26
Not completed — Condition under investigation worsened | 4 | 0 | 5 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 2
Not completed — Adverse Event | 1 | 2 | 0 | 3 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 28 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8931 160 mg bd | AZD8931 120 mg bd | AZD8931 80 mg bd | AZD8931 40 mg bd | AZD8931 40MG bd + Paclitaxel | Placebo + Paclitaxel | Total
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 94 | 96 | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at informed consent date
  Years
    Age for Part A | 52.7 (11.78) | 62.0 (16.97) | 47.2 (5.85) | 54.8 (11.07) | NA (NA) — Treatment in Part B only | NA (NA) — Treatment in Part B only | 52.6 (10.63)
    Age for Part B | NA (NA) — Treatment in Part A only | NA (NA) — Treatment in Part A only | NA (NA) — Treatment in Part A only | NA (NA) — Treatment in Part A only | 54.5 (11.87) | 53.1 (10.64) | 53.8 (11.26)
Age, Customized [Number; unit: Participants] — Age in years
  Participants
    < = 65 years | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | 72 | 84 | NA — Total not calculated because data are not available (NA) in one or more arms.
    > 65 years | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | 22 | 12 | NA — Total not calculated because data are not available (NA) in one or more arms.
    18 - <50 years | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | 34 | 38 | NA — Total not calculated because data are not available (NA) in one or more arms.
    50 - <=65 years | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | 38 | 46 | NA — Total not calculated because data are not available (NA) in one or more arms.
    >65 - <75 years | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | 18 | 11 | NA — Total not calculated because data are not available (NA) in one or more arms.
    >= 75 years | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | NA — Customized age tables were not presented for Part A | 4 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 4 | 94 | 96 | 206
  Male | 1 | 0 | 1 | 2 | 0 | 0 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Race: Black or African American | 0 | 0 | 0 | 0 | 4 | 1 | 5
  Race: Native Haiwaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: White | 6 | 2 | 6 | 6 | 75 | 74 | 169
  Race: Other | 0 | 0 | 0 | 0 | 13 | 18 | 31
  Race: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity: Hispanic or Latino | 6 | 2 | 6 | 6 | 35 | 31 | 86
  Ethnicity: Native American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Native Alaskan/Inuit | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: African | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: African-American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: African-Caribbean | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Ethnicity: Asian (other than Chinese and Japanese) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Ethnicity: Chinese | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Japanese | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Not Applicable | 0 | 0 | 0 | 0 | 47 | 49 | 96
  Ethnicity: Other | 0 | 0 | 0 | 0 | 12 | 14 | 26
  Ethnicity: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stratification: Prior taxane (This stratification information iis based on CRF data). [Number; unit: Participants] — Prior taxane in adjuvant setting
  Participants
    Prior taxane: Yes | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | 20 | 21 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Prior taxane: No | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | 74 | 75 | NA — Total not calculated because data are not available (NA) in one or more arms.
Stratification: Hormone receptor status (This stratification information iis based on CRF data). [Number; unit: Participants] — Hormone receptor status
  Participants
    Hormone receptor status Positive [ER+ and/or PgR+] | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | 76 | 75 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Hormone receptor status Negative [ER-/PgR-] | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | 18 | 21 | NA — Total not calculated because data are not available (NA) in one or more arms.
Stratification: Prior chemotherapy (This stratification information iis based on CRF data). [Number; unit: Participants] — Prior chemotherapy for locally advanced (not amenable to surgery) or metastatic breast cancer
  Participants
    Prior chemotherapy: Yes | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | 15 | 18 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Prior chemotherapy: No | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | NA — Not applicable for Part A | 79 | 78 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Phase I: The Number of Dose Limiting Toxicities in AZD8931 in Combination With Weekly Paclitaxel
Description: DLT is an AE or laboratory abnormality related to AZD8931, starting during the DLT evaluation period and meeting any of the following criteria (further detail in protocol): Symptomatic ocular surface lesion; CTCAE grade 4 haematological AE; CTCAE grade ≥3 of febrile neutropenia / neutropenia / thrombocytopenia / hyperkalaemia / hyperglycaemia / hypotension / urological toxicity / ILD / pneumonitis; QTcF interval > 500 msec, two ECGs ≥ 30 minutes apart; Symptomatic congestive cardiac failure and a drop in LVEF; Decrease in LVEF of ≥20% to below the LLN; CS rash remaining CTCAE grade ≥3 for ≥5 days despite optimal treatment; CTCAE grade ≥3 nausea, vomiting or diarrhoea, despite optimal therapy; Other CTCAE grade ≥3 toxicity which, in the opinion of the investigator, is CS and related to AZD8931; Delay to the administration of paclitaxel on D1 of Cycle 2 by ≥7 days. Patients could have more than one DLT.
Time Frame: Weekly visits for routine safety monitoring from Day 1 to Day 28 for each participant
Population: Safety population (all participants who received at least one dose)
Measure: Number; unit: Number of Dose Limiting Toxicities
Arm/Group | AZD8931 160 mg bd | AZD8931 120 mg bd | AZD8931 80 mg bd | AZD8931 40 mg bd
Number analyzed (Participants) | 6 | 2 | 6 | 6
Number of Dose Limiting Toxicities
  Total | 2 | 1 | 2 | 0
  Eye disorders: Keratitis | 1 | 0 | 0 | 0
  Eye disorders: Photophobia | 1 | 0 | 0 | 0
  Gastrointestinal disorders: Diarrhoea | 1 | 1 | 0 | 0
  Gastrointestinal disorders: Oesophagitis | 0 | 0 | 1 | 0
  Infections and infestations: Rash pustular | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: AZD8931 160 mg bd vs AZD8931 120 mg bd vs AZD8931 80 mg bd vs AZD8931 40 mg bd; A tolerated dose was defined as one where ≤25% of the patients experienced a DLT. If a dose was tolerated, an increased dose was to be investigated in another group of 3-6 evaluable patients. A non-tolerated dose was defined as one where >25% of the patients experience a DLT. If a dose was non tolerated, a decreased/intermediate dose could be investigated in another group of 3-6 evaluable patients. The maximum tolerated dose was determined as the maximum dose level that was defined as tolerated; Test type: Superiority or Other; Maximum Tolerated Dose = 40 — Dosing started at 160mg. Based on the data seen, 240mg with 33% patients with DLTs, 120mg with 50% patients with DLTs, 80mg with 33% of patients with DLTs and 40mg with 0% patients with DLTs, 40mg was deemed the maximum tolerated dose

2. Primary Outcome: Phase II: Progression-free-survival (PFS) Were Analyzed in Patients Treated With AZD8931 in Combination With Weekly Paclitaxel Versus Weekly Paclitaxel Alone
Description: Time from the date of randomization until the date of objective disease progression (as per RECIST 1.1) or the date of death (by any cause in the absence of progression)
Time Frame: Baseline and every 8 weeks, accessed up to data cut off on 11th April 2012
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Units Other Than Participants: events
Arm/Group | AZD8931 40MG bd + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 94 | 96
Number analyzed (events) | 69 | 68
Months | 8.7 [4.2 to 12.9] | 9.1 [3.4 to 14.8]
Statistical Analysis 1: Comparison: AZD8931 40MG bd + Paclitaxel vs Placebo + Paclitaxel; Originally, 166 patients were to be randomised to observe at least 133 progression events, based on HR=0.67, 80% power, 2-sided 5% significant level and a median of 6 months for the placebo arm. After 190 patients were randomised, the analysis was agreed to be performed at an similar level of maturity (70%) as originally planned (72%), after approximately 133 events; Test type: Superiority or Other; p = 0.679, Cox Proportional Hazard model — Statistical significance threshold at this analysis was 5%; Cox PH test with terms for treatment , prior taxane, hormone receptor status, prior chemotherapy for breast cancer and AZD8931 diagnostic test; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.76 to 1.52] — The Hazard Ratio is for AZD8931 40mg + paclitaxel / Placebo + paclitaxel, ie a hazard ratio <1 favours AZD8931 40mg + paclitaxel

3. Secondary Outcome: Phase II: Objective Tumour Response Rate (ORR) Was Compared in Patients Treated With AZD8931 in Combination With Weekly Paclitaxel Versus Weekly Paclitaxel Alone
Description: The number of subjects with at least one visit response of CR or PR (Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD), A ≥ 20% increase in the sum of diameters of target lesions and an absolute increase of ≥ 5mm; Stable disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Not Evaluable (NE), All target lesion measurements are missing or >1/3 target lesion measurements are missing and sum of diameters of non-missing target lesions does not qualify for PD; Not applicable (NA), No target lesions are recorded at baseline))
Time Frame: Baseline and every 8 weeks, accessed up to data cut off on 11th April 2012
Population: Evaluable for response set (EFR set is all FAS patients with measureable disease at baseline)
Measure: Number; unit: Participants
Arm/Group | AZD8931 40MG bd + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 88 | 85
Participants
  Total | 52 [4.2 to 12.9] | 35 [3.4 to 14.8]
  Complete Response | 11 | 6
  Partial Response | 41 | 29
Statistical Analysis 1: Comparison: AZD8931 40MG bd + Paclitaxel vs Placebo + Paclitaxel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.026, Logistic Regression — Statistical significance threshold at this analysis was 5%; Logistic reg. model with terms for treatment, prior taxane, hormone receptor status, prior chemotherapy for breast cancer and AZD8931 diagnostic test; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.09 to 3.75] — The odds Ratio is for AZD8931 40mg + paclitaxel / Placebo + paclitaxel, ie a odds ratio <1 favours AZD8931 40mg + paclitaxel

4. Secondary Outcome: Phase II: The Overall Survival (OS) Was Compared in Patients Treated With AZD8931 in Combination With Weekly Paclitaxel Versus Weekly Paclitaxel Alone
Description: The time from the date of randomization until the date of death due to any cause.
Time Frame: Weekly visits for routine safety monitoring, accessed up to data cut off on 11th April 2012
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Units Other Than Participants: events
Arm/Group | AZD8931 40MG bd + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 94 | 96
Number analyzed (events) | 28 | 24
Months | NA [13.1 to NA] — Median and the upper limit of the inter-quartile range for both treatment groups are not calculable due to an insufficient number of events | NA [14.1 to NA] — Median and the upper limit of the inter-quartile range for both treatment groups are not calculable due to an insufficient number of events
Statistical Analysis 1: Comparison: AZD8931 40MG bd + Paclitaxel vs Placebo + Paclitaxel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.607, Cox proportional hazard model — Statistical significance threshold at this analysis was 5%; Cox PH test with terms for treatment , prior taxane, hormone receptor status, prior chemotherapy for breast cancer; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.67 to 2.01] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: AEs will be collected from time of signed informed consent throughout the treatment period and including the 30-day safety follow up period after the last dose of study treatment
Description: In part B, SAEs considered related to study procedures should continue to be collected while patients are followed up for disease progression.
Arm/Group | AZD8931 40 mg bd | AZD8931 80 mg bd | AZD8931 120 mg bd | AZD8931 160 mg bd | AZD8931 40MG bd + Paclitaxel | Placebo + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/6 | 1/2 | 3/6 | 24/94 | 14/95
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 2/2 | 6/6 | 93/94 | 94/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8931 40 mg bd (N=6) | AZD8931 80 mg bd (N=6) | AZD8931 120 mg bd (N=2) | AZD8931 160 mg bd (N=6) | AZD8931 40MG bd + Paclitaxel (N=94) | Placebo + Paclitaxel (N=95)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST FIBROSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8931 40 mg bd (N=6) | AZD8931 80 mg bd (N=6) | AZD8931 120 mg bd (N=2) | AZD8931 160 mg bd (N=6) | AZD8931 40MG bd + Paclitaxel (N=94) | Placebo + Paclitaxel (N=95)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 23 (34) | 10 (14)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (27) | 5 (7)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 14 (42) | 39 (86)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ADDISON'S DISEASE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENOPIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLEPHARITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVAL DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 7 (7) | 5 (5)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 8 (8) | 3 (3)
ERYTHEMA OF EYELID (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EXOPHTHALMOS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXTRAOCULAR MUSCLE PARESIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EYE DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
EYE HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE PRURITUS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
EYELID OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
KERATITIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 1 (1)
MACULAR DEGENERATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOPIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
OCULAR TOXICITY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
PUNCTATE KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SCLERAL HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
XEROPHTHALMIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (9) | 12 (17)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 15 (20) | 7 (11)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ANAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAL PRURITUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
CHAPPED LIPS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (8) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 19 (25) | 23 (29)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 5 (12) | 6 (25) | 2 (3) | 5 (15) | 78 (247) | 33 (65)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (19) | 9 (9)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GINGIVITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GLOSSITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GLOSSODYNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (4)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIP DRY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIP PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUCOUS STOOLS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (5) | 39 (69) | 30 (39)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL DYSAESTHESIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ORAL MUCOSAL BLISTERING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL TOXICITY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PERIANAL ERYTHEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
RECTAL FISSURE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 3 (7) | 1 (1) | 1 (1) | 20 (26) | 3 (3)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (8)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 24 (43) | 14 (27)
ASTHENIA (General disorders) | 5 (8) | 6 (11) | 2 (2) | 5 (7) | 25 (30) | 12 (16)
AXILLARY PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATHETER SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 25 (40) | 25 (29)
FEELING COLD (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
INFUSION SITE DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IRRITABILITY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MUCOSAL DRYNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 21 (35) | 9 (9)
NODULE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 11 (18)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (16) | 4 (17)
PYREXIA (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 7 (9) | 11 (11)
SPINAL PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
XEROSIS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GALLBLADDER PAIN (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (4)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 9 (11) | 3 (3)
DERMATOPHYTOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HORDEOLUM (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAIL BED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 9 (12)
ONYCHOMYCOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ORAL PUSTULE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 24 (30) | 5 (6)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PHARYNGOTONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 14 (18) | 2 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 6 (9)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRACHEITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (11) | 11 (13)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 19 (29) | 13 (22)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
VULVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESCHAR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECALL PHENOMENON (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SKIN INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAPILLARY FRAGILITY TEST (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM CHANGE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 4 (5)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
PULMONARY PHYSICAL EXAMINATION ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINE COLOUR ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 3 (3)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 5 (13)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (11) | 2 (2)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 5 (6)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 14 (25) | 19 (26)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (20) | 16 (30)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 2 (3)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (5)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 7 (7)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 11 (14)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 9 (9)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (19) | 16 (25)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ANOSMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHONIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 7 (10) | 7 (10)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 9 (13) | 2 (2)
FACIAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 13 (21) | 16 (18)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4)
HYPOGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPOKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOSMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 4 (4)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MOTOR DYSFUNCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 28 (34) | 25 (27)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (18) | 19 (22)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (13) | 11 (13)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AFFECT LABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 11 (13)
APATHY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRADYPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (4)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (13) | 14 (14)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
NERVOUSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLADDER PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 3 (4)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
BREAST DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST ENGORGEMENT (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST INFLAMMATION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
GENITAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GENITAL RASH (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL INFLAMMATION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
VULVAL ULCERATION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VULVOVAGINAL BURNING SENSATION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 0 (0) | 2 (2) | 12 (14) | 19 (26)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 7 (10) | 8 (8)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 19 (21) | 11 (12)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPEROXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINALGIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 45 (45) | 48 (49)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (40) | 2 (2)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 2 (2)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HEAT RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MADAROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 7 (7) | 8 (8)
NAIL DYSTROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
NAIL PIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 18 (19) | 6 (6)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (5) | 5 (19) | 1 (1) | 4 (15) | 59 (136) | 20 (26)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SKIN CHAPPED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN PLAQUE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SKIN STRIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 2 (5)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
HYPERAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 7 (24) | 3 (4)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
TINEA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URETERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (2) | 2 (3) | 21 (27) | 15 (17)
FLUID RETENTION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROTOXICITY (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 5 (8) | 10 (19)
INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEUKOCYTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (5)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 32 (36) | 7 (7)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. The primary statistical analysis of PFS was performed, but the planned analyses of overall survival at 50% maturity, and of PFS at 50% OS maturity, were not performed.
2. AEs were coded using MedDRA v14.0 (part A) and MedDRA v15.0 (part B).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days